CLINICAL TRIAL: NCT04531137
Title: Conjugated Linoleic Acid Combined With Nutrition Counseling Consequences on Body Weight and Body Fat Mass in Overweight and Obese Adult
Brief Title: Conjugated Linoleic Acid on Body Weight and Body Fat Mass for 12 Weeks
Acronym: CLAPSProject
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Indonesia University (Other)
Collaborators: BASF (Industry)
Responsible Party: Principal Investigator, Fiastuti Witjaksono, Principal Investigator, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 19-10-1189
Record Dates: First submitted 2020-08-11; First posted 2020-08-28 (Actual); Last update posted 2021-08-17 (Actual); Status verified 2021-08

CONDITIONS: Overweight and Obesity; Body Weight
Keywords: conjugated linoleic acid; body fat mass; body composition; nutrition counseling
MeSH Terms: conditions — Overweight; Obesity; Body Weight

STUDY DESIGN:
Intervention Model Description: This study consists of intervention and control groups. The intervention group will receive CLA-fortified milk powder containing 3.4 gram CLA for one a day. The control group will receive milk powder for one a day. In each group, the intervention phase will be conducted in 12 weeks. Each group will also receive nutritional counseling and nutrition module
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CLA-fortified milk powder (Experimental): Respondents will receive CLA-fortified milk powder containing 3.4 gram for one a day for 12 weeks. They will also receive individualized nutrition counseling and nutrition module at weeks 0, 4, and 8.
  Interventions: Dietary Supplement: CLA-fortified milk powder; Other: Nutrition Counseling
- Placebo (Other): Respondents will receive a placebo milk powder for one a day for 12 weeks. They will also receive individualized nutrition counseling and nutrition module at weeks 0, 4, and 8.
  Interventions: Other: Placebo; Other: Nutrition Counseling

INTERVENTIONS:
Dietary Supplement: CLA-fortified milk powder — 3.4 gram of CLA-fortified milk powder one a day for 12 weeks
  Arms: CLA-fortified milk powder
Other: Placebo — Placebo milk powder one a day for 12 weeks
  Arms: Placebo
Other: Nutrition Counseling — Individualized nutrition counseling using nutrition module at week 0, 4, and 8 for 30-45 minutes each session

SUMMARY:
This study has purpose to assess the effect of conjugated linoleic acid (CLA)-fortified milk powder with nutrition counseling and nutrition module in body weight and body fat mass among overweight and obese adult in Indonesia

DETAILED DESCRIPTION:
After being informed of the potential benefits and risks regarding the study, the respondents were asked to sign the consent. The respondents who met the criteria of overweight/ obese without any historical diseases will be randomized into intervention or placebo groups. The intervention will be given for 12 weeks (CLA-fortified milk powder 3.4 gram, once-daily consumption). Both the intervention and placebo groups will also receive nutrition counseling and nutrition module.

ELIGIBILITY:
Inclusion Criteria:

1. Body mass index (BMI) 23 - 24.9 kg/m2 for overweight and ≥ 25 kg/m2 for obese
2. Fat mass percentage (FM%) of ≥ 20% for men and ≥ 30% for women
3. Agree to follow the study

Exclusion Criteria:

1. Lactose intolerance
2. Undergoing treatment (e.g., antibiotics and/or anti-inflammatory or immunosuppressant drugs and weight loss)
3. Any physical condition that might be contraindicated to dietary restrictions
4. Any non-communicable disease (e.g., Diabetes Mellitus, Chronic Kidney Disease, Cancer, Hypertension)
5. Pregnant

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 84 (Estimated)
Dates: Start 2020-08-05 (Actual); Primary Completion 2021-11 (Estimated); Study Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
Change of body weight | Baseline (after signing the consent) week-0, week-4, week-8, and week-12 (endline)
  to investigate the change of body weight before, during and after intervention. Using Seca® type 876 is calibrated scale to the nearest 0.1 kilogram. The lower body weight indicates better outcome
Change of body fat mass | Baseline (after signing the consent) week-0 and week-12 (endline)
  to investigate the change of body fat mass before and after intervention. Using Dual-energy X-ray absorptiometry (DXA GE Lunar® Prodigy 64179). The lower body fat mass indicates better outcome
Change of body fat mass | Baseline (after signing the consent) week-0, week-4, week-8, and week-12 (endline)
  to investigate the change of body fat mass before, during, and after intervention. Using Bod Pod (Cosmed®). The lower body fat mass indicates better outcome

SECONDARY OUTCOMES:
Change of Waist hip ratio | Baseline (after signing the consent) week-0, week-4, week-8, and week-12 (endline)
  to investigate the change of waist hip ratio before, during, and after intervention. Waist hip ratio is obtained by dividing the waist circumference and hip circumference. Tape measurement (Seca® type 201) is calibrated scale to nearest 0.1 centimeter. The lower body fat mass indicates better outcome
Change of Low Density Lipoprotein (LDL) | Baseline (after signing the consent) week-0 and week-12 (endline)
  to investigate the change of low density lipoprotein (LDL) in miligram per deciliter before and after intervention. The lower change of LDL indicates the better outcome. Enzymatic method
Change of High Density Lipoprotein (HDL) | Baseline (after signing the consent) week-0 and week-12 (endline)
  to investigate the change of high density lipoprotein (HDL) in miligram per deciliter before and after intervention. The higher change of HDL indicates the better outcome. Enzymatic method
Change of Total of Cholesterol | Baseline (after signing the consent) week-0 and week-12 (endline)
  to investigate the change of total of cholesterol in miligram per deciliter before and after intervention. The lower change of total of cholesterol indicates the better outcome. Enzymatic method
Change of Triglyceride | Baseline (after signing the consent) week-0 and week-12 (endline)
  to investigate the change of triglyceride in miligram per deciliter before and after intervention. The lower change of triglyceride indicates the better outcome. Enzymatic method
Dietary intake (semi quantitative food frequency questionnaire) | Baseline (after signing the consent) week-0, week-8 and week-12 (endline)
  to investigate the dietary intake before, during, and after intervention using semi quantitative food frequency questionnaire. The higher number of dietary intake indicates the better outcome
Dietary intake (24-hours recall) | Baseline (after signing the consent) week-0, week-8 and week-12 (endline)
  to investigate the dietary intake before, during, and after intervention using 24-hours recall. The higher dietary intake indicates the better outcome
Change of knowledge | Baseline (after signing the consent) week-0 and week-12 (endline)
  to investigate the score of knowledge before and after the intervention. Using validated questionnaire of knowledge. Minimum score is 0 and maximum score is 100.The higher score of knowledge after intervention indicates the better outcome.
Change of attitude | Baseline (after signing the consent) week-0 and week-12 (endline)
  to investigate the score of attitude before and after the intervention. Using validated questionnaire of attitude. Minimum score is 0, maximum score is 100. The higher score of attitude after intervention indicates the better outcome.
Physical activity level | Baseline (after signing the consent) week-0, week-4, week-8, and week-12 (endline)
  to investigate the physical activity level before, during and after intervention. Using International Physical Activity Questionnaire. The category of physical activity level are low (<600 metabolic equivalents), moderate (>=600 - 3000 metabolic equivalents) and high (>=3000 metabolic equivalents).

CONTACTS AND LOCATIONS:
Overall Officials: Fiastuti Witjaksono, Doctoral, Principal Investigator — Department of Nutrition, Faculty of Medicine of Universitas Indonesia
Locations (1):
- Faculty of Medicine Universitas Indonesia, Jakarta Pusat, Jakarta Special Capital Region, Indonesia

IPD SHARING:
Plan to Share IPD: No